

# Protocol for: Neonatal resuscitation: comparing sustained inflations to standard practice

A prospective randomised controlled trial assessing the efficacy of sustained inflations in neonatal resuscitation compared to repeated shorter inflation breaths

#### Sponsor

Sponsoring Organisation/s: King's College London and King's College Hospital NHS

Name of Sponsor Representative: Keith Brennan, Director of Research Management & Director of Administration (Health Schools)

Address: Room 1.8 Hodgkin Building, Guy's Campus, King's College London, LONDON, SE1 4UL.

Tel: 020 7848 6960

Email: keith.brennan@kcl.ac.uk

Name of Sponsor Representative: Liba Stones, R&D Manager,

Address: King's College Hospital, 161 Denmark Hill, London, SE5 8EF,

Tel: 020 3299 3841

e-mail: liba.stones@nhs.net

#### **Chief Investigator**

Name: Professor Anne Greenough

Address: 4th Floor Golden Jubilee Wing, King's College Hospital, Denmark Hill, SE5

9RS

Tel: 020 3299 3037

Email: anne.greenough@kcl.ac.uk

#### Name and address of Investigator(s)

Name: Dr Katie Hunt

Address: 4th Floor Golden Jubilee Wing, King's College Hospital, Denmark Hill, SE5

9RS

Tel: 020 3299 4564

Email: katie.a.hunt@kcl.ac.uk

#### Statistician

Name: Professor Anne Greenough

Address: 4th Floor Golden Jubilee Wing, King's College Hospital, Denmark Hill, SE5

9RS

Tel: 020 3299 3037

Email: anne.greenough@kcl.ac.uk

#### 2 Trial Objectives, Design and Statistics

- 2.1. Trial Objectives
- 2.2 Trial Design & Flowchart
- 2.3 Trial Flowchart
- 2.4 Trial Statistics

## 3. Sample Size, Selection and Withdrawal of Subjects

- 3.1 Inclusion
- 3.2 Exclusion
- 3.3 Criteria for Premature Withdrawal

#### 4. Study procedures

- 4.1 Screening Procedures
- 4.2 Randomisation Procedures
- 4.3 Schedule of Treatment for each visit
- 4.4 Follow up procedures
- 4.5 Radiology assessments
- 4.6 End of Study Definition

#### 5. Laboratories

- 5.1 Central/local Laboratories
- 5.2 Sample collection/labelling logging
- 5.3 Sample analysis procedures
- 5.4 Sample storage procedures
- 5.5 data Recording/Reporting
- 5.6 Sample receipt/chain of custody/Accountability
- 5.7 Tissue Sample Transfer

#### 6. Assessment of Safety

- 6.1 Ethics Reporting
- 7. Trial Steering Committee
- 8. Direct Access to Source Data and Documents
- 9. Ethics & Regulatory Approvals

#### 10. Data Handling

- 10.1 Case Report From
- 10.2 Record retention and Archiving
- 10.3 Compliance
- 10.4 Clinical Governance issues
- 10.4 Non Compliance

#### 11. Finance & Publication Policy

# **Study Synopsis**

| Title | Neonatal resuscitation: comparing sustained inflations to repeated shorter inflation breaths |
|---|---|
| Protocol Short Title/Acronym | Neonatal Resuscitation: sustained inflation |
| Protocol Version number and Date | 4 11/1/18 |
| Study Phase if not mentioned in title | |
| Is the study a Pilot? | No |
| Study Duration | 12 months |
| Methodology | Randomised controlled trial |
| Sponsor name | Mr Keith Brennan/Ms Liba Stones |
| Chief Investigator | Professor Anne Greenough |
| REC number | 16 LO 1718 |
| Medical condition or disease under investigation | Need for resuscitation at delivery in babies born prematurely |
| Purpose of clinical trial | To assess whether 15 second inflations are more effective at stimulating spontaneous breathing than five shorter inflation breaths of 2-3 seconds. |
| Primary objective | To assess whether sustained inflations provoke active inflations sooner during resuscitation than repeated shorter inflation breaths |
| Secondary objective (s) | To assess whether sustained inflations improve tidal volume exchange and end tidal carbon dioxide levels compared to repeated shorter inflation breaths, and to collect data regarding any adverse outcomes. |
| Number of Subjects/Patients | 48 + |
| Trial Design | Randomised controlled trial |
| Endpoints | Equal distribution of gestational age between groups |
| Main Inclusion Criteria | Any baby born <34/40 requiring resuscitation at delivery |
| Statistical Methodology and Analysis | Non-parametric statistics |

## Glossary of Terms and Abbreviations

AE Adverse Event

AR Adverse Reaction

ASR Annual Safety Report
CA Competent Authority
CI Chief Investigator

CRF Case Report Form

CRO Contract Research Organisation

DMC Data Monitoring Committee

EC European Commission

GAFREC Governance Arrangements for NHS Research Ethics Committees

ICF Informed Consent Form

ISRCTN International Standard Randomised Controlled Trial Number

MA Marketing Authorisation

MS Member State

Main REC Main Research Ethics Committee

NHS R&D National Health Service Research & Development

PI Principle Investigator
QA Quality Assurance

QC Quality Control

Participant An individual who takes part in a clinical trial

RCT Randomised Controlled Trial
REC Research Ethics Committee

SAE Serious Adverse Event

SDV Source Document Verification
SOP Standard Operating Procedure

SSA Site Specific Assessment
TMG Trial Management Group
TSC Trial Steering Committee

#### 1. Introduction

Around 10% of newborns will require some form of assistance after delivery, with babies born more prematurely more likely to require resuscitation.<sup>1</sup>

Current UK guidelines advise initial resuscitation with the delivery of five 'inflation breaths' lasting 2-3 seconds with peak inflation pressure of 30cmH2O (20-25cm H2O in premature neonates).<sup>2</sup> Previous studies have shown that despite resuscitation training, clinicians in both simulated and real resuscitation scenarios do not deliver the recommended duration of inflation breaths<sup>3</sup>. This, combined with leaks around the facemask often being as large as 50% or greater, contributes to low expired tidal volumes during resuscitation, thus increasing the likelihood of hypoxia and delay in establishing effective respiration.

The use of sustained inflations (up to 15 seconds), rather than intermittent shorter inflation breaths, has shown promising results, with reduction in the need for intubation, and the need for and duration of mechanical ventilation.<sup>4–7</sup> Around 30% of units in Germany use sustained inflations as first line delivery room management, as do many other hospitals around the world.<sup>8</sup> Resuscitation guidelines from the USA, UK and Europe suggest that sustained inflations should be researched further.<sup>9,10</sup>

Several studies have shown that for several lengths of inflation breaths, the expired tidal volume achieved is higher if the baby makes respiratory effort during the inflation (active inflation),<sup>3,11,12</sup> and that stimulation of spontaneous respiratory effort is a key part in establishing an FRC, enabling spontaneous breathing, and increasing the likelihood of successful resuscitation.

To date, there are no studies directly comparing whether prolonged inflations are more successful at provoking an inspiration than other methods of resuscitation. We therefore aim to compare a 15 second sustained inflation to repeated shorter inflations to determine which is more effective.

- 1. Aziz K, Chadwick M, Baker M, Andrews W. Ante- and intra-partum factors that predict increased need for neonatal resuscitation. *Resuscitation*. 2008;79(3):444-452. doi:10.1016/j.resuscitation.2008.08.004.
- 2. (UK) RC. NLS Guidelines (Resuscitation council). resus.org.uk.
- 3. Murthy V, Dattani N, Peacock JL, et al. The first five inflations during resuscitation of prematurely born infants. *Arch Dis Child Fetal Neonatal Ed*. 2012;97(4):F249-F253. doi:10.1136/archdischild-2011-300117.
- 4. te Pas AB, Walther FJ. A Randomized, Controlled Trial of Delivery-Room Respiratory Management in Very Preterm Infants. *Pediatrics*. 2007;120(2):322-329. doi:10.1542/peds.2007-0114.
- 5. Grasso C, Sciacca P, Giacchi V, et al. Effects of Sustained Lung Inflation, a lung recruitment maneuver in primary acute respiratory distress syndrome, in respiratory and cerebral outcomes in preterm infants. *Early Hum Dev.* 2015;91(1):71-75. doi:10.1016/j.earlhumdev.2014.12.002.
- 6. Lista G, Boni L, Scopesi F, et al. Sustained Lung Inflation at Birth for Preterm Infants: A Randomized Clinical Trial. *Pediatrics*. 2015;135(2):e457-e464. doi:10.1542/peds.2014-1692.
- 7. El-Chimi MS, Awad HA, El-Gammasy TM, El-Farghali OG, Sallam MT, Shinkar DM. Sustained vs. Intermittent Lung Inflation for Resuscitation of Preterm Infants: a

- Randomized Controlled Trial. *J Matern Neonatal Med*. July 2016:1-21. doi:10.1080/14767058.2016.1210598.
- 8. Fuchs H. German experience in the management of ELGAN infants. *Acta Biomed*. 2015;86 Suppl 1:16-20. http://www.ncbi.nlm.nih.gov/pubmed/26135950. Accessed July 21, 2016.
- 9. Wyllie J, Ainsworth S. What is new in the European and UK neonatal resuscitation guidance? *Arch Dis Child Fetal Neonatal Ed*. April 2016:fetalneonatal 2015-309472. doi:10.1136/archdischild-2015-309472.
- Wyckoff MH, Aziz K, Escobedo MB, et al. Part 13: Neonatal Resuscitation: 2015
   American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015;132(18 Suppl 2):S543-S560. doi:10.1161/CIR.000000000000000267.
- 11. Schilleman K, van der Pot CJMM, Hooper SB, Lopriore E, Walther FJ, te Pas AB. Evaluating Manual Inflations and Breathing during Mask Ventilation in Preterm Infants at Birth. *J Pediatr*. 2013;162(3):457-463. doi:10.1016/j.jpeds.2012.09.036.
- 12. van Vonderen JJ, Hooper SB, Hummler HD, Lopriore E, te Pas AB. Effects of a Sustained Inflation in Preterm Infants at Birth. *J Pediatr*. 2014;165(5):903-908.e1. doi:10.1016/j.jpeds.2014.06.007.

## 2 Trial Objectives, Design and Statistics

## 2.1. Trial Objectives

To assess whether a 15 second inflation are more effective at stimulating spontaneous breathing than five shorter breaths of 2-3 seconds, evidenced by a greater number of active inflations and superior tidal volume exchange and end tidal carbon dioxide levels.

#### 2.2 Trial Design & Flowchart

Randomised controlled trial.

#### 2.3 Trial Flowchart



## 3. Sample Size, Selection and Withdrawal of Subjects

We have previously demonstrated that active compared to passive inflations during resuscitation at least double expiratory tidal volumes and end tidal CO2 levels. (An active inflation is one where the baby makes inspiratory effort during a mechanical inflation.) During resuscitation with short inflations, all infants had an active inflation by 50 seconds, but the active inflation occurred earlier in those who received longer rather than shorter mechanical inflations. We therefore postulate that over the first minute of resuscitation the total expiratory tidal volume (minute volume) will be 25% higher in the prolonged inflation group. Randomisation of 40 infants will allow us to detect one standardised difference in the minute volume between the two groups with 90% power at the 5% level. The standard deviation in our previous cohort in minute volume was 71mls/min/kg, that is 25% of the maximum minute volume achieved in our previous cohort.

At reaching the prespecified sample size we have a two week discrepancy in gestational age between the two groups, and therefore we will continue to recruit to the study until this is balanced. We anticipate that around 60 infants will be required but this will be reviewed after every 4 babies to be recruited.

#### **Inclusion Criteria**

Infants born less than 34 weeks of gestation requiring resuscitation at delivery.

#### **Exclusion Criteria**

Major congenital abnormalities

#### **Criteria for Premature Withdrawal**

Withdrawal of parental consent

## 4. Study procedures

#### **Informed Consent Procedures**

Preterm delivery may often occur without significant prior warning. When women are in preterm labour, it may be inappropriate to approach them regarding research at this potentially distressing time, particularly as this may be very close to the point of delivery. We therefore intend to conduct this study as emergency research without prior informed consent, and will approach parents as soon as is practical after delivery to explain the research and to gain consent for analysis of resuscitation data and collection of further data. Information will be displayed on the antenatal wards regarding research without prior consent and contact details if any parents wish to discuss this.

#### 4.1 Screening Procedures

There are no study specific screening procedures prior to entry into the study.

#### 4.2 Randomisation Procedures

A random number generator will be used and allocations concealed in sealed opaque envelopes, opened immediately when it is deemed that resuscitation is required.

#### 4.3 Schedule of Events for each visit

Infants randomised to the routine care group will receive resuscitation as per NLS protocols, with the addition of respiratory function monitoring. Infants randomised to the sustained inflation group will receive a 15 second sustained inflation at 25cmH<sub>2</sub>O in place of the five inflation breaths and this will be repeated in situations where, under normal circumstances, the five inflation breaths would be repeated (e.g. no chest rise seen.) The decision to initially resuscitate via facemask or to immediately intubate will be taken on usual clinical grounds, as will any subsequent decisions to intubate, perform chest compressions, or deliver medications. Resuscitation will otherwise proceed as per normal practice and, as above, the decision to intubate etc will be taken on normal clinical grounds by the team performing the resuscitation.

#### 4.4 Follow up Procedures

Data regarding rates of pneumothorax, patent ductus arteriosus, intraventricular haemorrhage, need for mechanical ventilation in the first 72 hours of life, and mortality will be recorded.

## 4.5 Radiology Assessments (not applicable)

Not applicable

## 4.6 End of Study Definition

Following completion of the measurements and analysis of the results of the required number of infants, the REC will be informed that the study has been completed.

## 5. Laboratories (not applicable)

## 6. Assessment of Safety

Some studies have shown small, non-significant trends towards increased incidence of pneumothorax and intraventricular haemorrhage with sustained inflations. Another trial has shown a reduction in the incidence of air leak with sustained inflation, and animal studies have demonstrated improved stabilisation of cerebral blood flow with sustained inflation. Meta-analysis of four trials has shown an increase in the occurrence of patent ductus arteriosus requiring treatment, but these trials were heterogenous in terms of the oxygen concentration used and length and pressure of sustained inflation. Sustained inflations have not previously been compared to five shorter inflation breaths lasting 2-3 seconds. Sustained inflations are used as a routine standard of care in many hospitals worldwide.

#### 6.1 Ethics Reporting

Reports of related and unexpected serious adverse events will be submitted to the Main REC within 15 days of the chief investigator becoming aware of the event, using the NRES template. The parents will be informed of any events as soon as possible and be provided with an opportunity to meet with clinical and research team. The results of any reports or investigations relating to the events will also be communicated to the parents in writing.

## 7. Trial Steering Committee

#### 8. Ethics & Regulatory Approvals

We will make an application via IRAS for HRA and NHS REC review and approval.

#### Confidentiality

Analysis of the data will take place at King's College Hospital and is to be undertaken by a clinical research fellow and by Professor Greenough, the chief investigator.

Each patient will be assigned a unique patient identifier, under which patient data will be anonymously stored on a password protected computer. All paper copies containing patient identifiable data will be kept in a locked filing cabinet until the patients are 25 years of age. Only the principal investigator and research fellow involved in the study will have access to the data, the principal investigator will act as custodian.

#### **Case Report Form**

Elements included in each case report form (CRF):

- -Unique patient identifier
- -Date of parental consent

- -Eligibility criteria checklist
- -Date of resuscitation
- -Any adverse events noted

Completion of the CRF will be the responsibility of the clinical research fellow.

## **Record Retention and Archiving**

Records will be held in a locked filing cabinet located within the research office based at the neonatal unit of Kings College Hospital. Access is limited to the clinical research fellow and Chief Investigator.

## Compliance

The CI will ensure that the trial is conducted in compliance with the principles of the Declaration of Helsinki (1996), and in accordance with all applicable regulatory requirements including but not limited to the Research Governance Framework, Trust and Research Office policies and procedures and any subsequent amendments.

#### **Clinical Governance Issues**

#### -Audit and Inspection

Accurate records of all research activity including copies of the consent forms and completed case report forms will be safely stored and audited for compliance if requested.

#### -Non-Compliance

The sponsor will maintain a log of the non-compliances to ascertain if there are any trends developing which to be escalated. The sponsor will assess the non-compliances and action a timeframe in which they need to be dealt with. Each action will be given a different timeframe dependant on the severity. If the actions are not dealt with accordingly, the R&D Office will agree an appropriate action, including an on-site audit.

## 10. Finance and Publication Policy

Appendix 1 – Information with regards to Safety Reporting in Non-CTIMP Research

| Appendix 1 - Information with regards to Safety Reporting in Non-Crimin Research | | | | |
|---|---|---|---|---|
| | Who | When | How | To Whom |
| SAE | Chief<br>Investigator | -Report to Sponsor within 24 hours of learning of the event -Report to the MREC within 15 days of learning of the event | SAE Report form for Non-<br>CTIMPs, available from<br>NRES website. | Sponsor and<br>MREC |
| Urgent Safety<br>Measures | Chief<br>Investigator | Contact the Sponsor<br>and MREC<br>Immediately<br>Within 3 days | By phone Substantial amendment | Main REC and Sponsor Main REC with a |

| | | | form giving notice in writing setting out the reasons for the urgent safety measures and the plan for future action. | copy also sent to<br>the sponsor. The<br>MREC will<br>acknowledge this<br>within 30 days of<br>receipt. |
|---|---|---|---|---|
| <u>Progress</u><br><u>Reports</u> | Chief<br>Investigator | Annually ( starting 12 months after the date of favourable opinion) | Annual Progress Report<br>Form (non-CTIMPs)<br>available from the NRES<br>website | Main REC |
| Declaration of the conclusion or early termination of the study | Chief<br>Investigator | Within 90 days (conclusion) Within 15 days (early termination) The end of study should be defined in the protocol | End of Study Declaration form available from the NRES website | Main REC with a copy to be sent to the sponsor |
| Summary of final Report | Chief<br>Investigator | Within one year of<br>conclusion of the<br>Research | No Standard Format However, the following Information should be included:- Where the study has met its objectives, the main findings and arrangements for publication or dissemination including feedback to participants | Main REC with a copy to be sent to the sponsor |